CLINICAL TRIAL: NCT00502177
Title: Quality of Life Study for Pediatric and Adult Patients Undergoing Hyperthermic Peritoneal Perfusion With Cisplatin
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-1106
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Peritoneal Neoplasms
Keywords: Continuous Hyperthermic Peritoneal Perfusion; Peritoneal Neoplasms; Quality of Life; Questionnaire; Survey; CHPP
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Quality of Life Questionnaire: Patients undergoing continuous hyperthermic peritoneal perfusion with cisplatin and their parents/caregivers.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — QOL Questionnaires taking a total of 10 minutes to complete.
  Other Names: Survey

SUMMARY:
Objectives:

The overall objective of this prospective study is to provide a descriptive analysis of the quality of life of cancer patients enrolled on M. D. Anderson Cancer Center Protocol 2009-0528, "A Phase II Study of Hyperthermic Peritoneal Perfusion (HIPEC) for Adolescent and Young Adults with Desmoplastic Small Round Cell Tumor (DSRCT) and Other Non-carcinomas".

Specific Aim 1: To examine the quality of life of patients who undergo HIPEC longitudinally. It is hypothesized that physical health and functioning concerns, as reported by parent/child dyads on the Pediatric Quality of Life Cancer Module Version 3.0 (PedsQL) and the PedsQL 4.0 Generic Core Scales, will will remain stable or improve, following the surgical procedures and peritoneal perfusion described in Protocol 2009-0528.

Specific Aim 2: To assess parent and patient perception of the relative benefit of HIPEC longitudinally. It is hypothesized that parents and patients will perceive HIPEC to be beneficial across time, despite the temporary postoperative pain and discomfort that is associated with the procedure. This will be done by means of a non-validated question that is specific to the surgery.

Exploratory Aim: To determine whether quality of life following HIPEC varies by demographic factors (e.g., age, culture), intraoperative cisplatin dose level, or subsequent treatment modalities. Some patients who undergo HIPEC might subsequently be treated with other Phase II chemotherapy agents and/or palliative radiation, and comparing quality of life in these subgroups will be of value. Also the quality of life for groups of patients enrolled in Protocol 2009-0528 at each intraoperative cisplatin dose level will be compared.

DETAILED DESCRIPTION:
Child Participant:

Study Participation:

If you agree to take part in this study, you will complete questionnaires about your quality of life. If you do not want to participate in this study, your parent or caregiver may still participate and complete the parent/caregiver questionnaires if he/she chooses.

The questionnaires will ask about your experiences with pain, nausea, anxiety, worry, thinking and reasoning ability, physical appearance, communication, and your emotional, social, school, and physical functioning. Both questionnaires should take about 10 minutes to complete in total, or longer if you need more time. You will also be asked about whether you worry about the surgery being effective.

If you are 4 years old or younger, your parent/caregiver will fill out the questionnaires for you.

If you are between 5 and 7 years old, the interviewer will go over the questionnaires with you.

If you are between 8 and 18 years old, you will fill out the questionnaires on your own.

The questionnaires will be filled out in the week before the surgery, 1 month after the surgery, 3 months and 6 months after the surgery.

You will only come in if you already have a scheduled visit because of the study you are presently on. However, if you are no longer on that study then you will still be asked to complete the questionnaires at the 1, 3 and 6-month time points. This can be done by telephone or at other regularly scheduled visits at those time points.

Length of Study:

Your participation in this study will be over after you finish the 6-month questionnaires.

This is an investigational study. Up to 20 parents and 20 children will participate in this study. All will be enrolled at M. D. Anderson.

Parent/Caregiver Participant:

Parent Participation:

If you agree to take part in this study, you will complete questionnaires about your perception of your child's quality of life. If your child does not want to participate in this study, you may still participate and complete the parent/caregiver questionnaire, if you so choose. If your child is too ill to participate in this study, you will not be asked to complete his/her questionnaires on his/her behalf.

The questionnaires will ask about your child's quality of life regarding pain, nausea, anxiety, worry, cognitive functioning (thinking and reasoning), physical appearance, communication, and his or her emotional, social, school, and physical functioning. Both questionnaires should take about 10 minutes to complete in total.

You will also be asked a surgery-specific question about whether your child worries about the effectiveness of the surgery.

Length of Study:

Your participation in this study will be over after completion of the 6-month questionnaires.

This is an investigational study. Up to 20 parents and 20 children will participate in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria

1. All participants must be English or Spanish speaking.
2. A patient enrolled on Protocol 2009-0528, and/or one parent or adult non-parent primary caretaker of the child enrolled on Protocol 2009-0528.
3. Patients greater than or equal to 1 year.

Exclusion Criteria:

1. Patients not enrolled on Protocol 2009-0528 will be excluded from this study.
2. Patients less than 1 year.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients undergoing continuous hyperthermic peritoneal perfusion with cisplatin and their parents/caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2007-06-19 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
PedsQL 4.0 Generic Core Scale | 6 Months
  The mean change in PedsQL 4.0 Generic Core Total Score over time (i.e., prior to operation vs. 6-months post-operation. The PedsQL 4.0 Generic Core will be administered to each child to ascertain their quality of life at the two time points).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Hayes-Jordan, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org